CLINICAL TRIAL: NCT07004790
Title: Prognostic Value of Transcranial Doppler Ultrasound in the Clinical Evolution of Patients With Acute Ischemic Stroke: A Prospective Observational Study
Brief Title: Prognostic Value of Transcranial Doppler Ultrasound in the Clinical Evolution of Patients With Acute Ischemic Stroke. The TRADE-AIS Study
Acronym: TRADE-AIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jose Ivan Rodriguez de Molina Serrano (Other)
Responsible Party: Sponsor-Investigator, Jose Ivan Rodriguez de Molina Serrano, Head of Research and Medical Education Clinica Mexico, Clinica Mexico
Organization: Clinica Mexico (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CMX0004
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stroke
Keywords: stroke; transcranial doppler; Prognosis; Middle Cerebral Artery; Cerebral Hemodynamics; Mexico
MeSH Terms: conditions — Stroke | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Intervention Model Description: Participants with confirmed acute ischemic stroke will be enrolled consecutively and followed as a single cohort. All participants will undergo baseline clinical assessment and transcranial Doppler ultrasound within 24 hours of symptom onset. No grouping or randomization will be applied. The study will observe natural clinical progression and outcomes without intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inpatient Stroke confirmed (Other): All participants diagnosed with acute ischemic stroke will undergo standard clinical evaluation and transcranial Doppler ultrasound within 24 hours of symptom onset. No interventions are assigned by the study. Clinical and hemodynamic data will be collected to assess prognostic associations with short-term outcomes. All patients are managed according to routine care protocols determined by the attending medical team.
  Interventions: Diagnostic Test: Transcranial Doppler Ultrasound

INTERVENTIONS:
Diagnostic Test: Transcranial Doppler Ultrasound — A non-invasive bedside diagnostic procedure used to measure cerebral blood flow velocities and pulsatility index in intracranial arteries, primarily the middle cerebral artery (MCA). The test is performed within the first 24 hours of symptom onset using standard ultrasound equipment with a 2-MHz probe. The data collected is used solely for prognostic evaluation and does not influence treatment decisions.

SUMMARY:
This prospective observational study aims to determine whether specific parameters measured by transcranial Doppler ultrasound (TCD) can predict clinical outcomes in patients with acute ischemic stroke (AIS). The primary objective is to evaluate the association between middle cerebral artery (MCA) flow velocities and short-term neurological improvement. Secondary outcomes include the presence of collateral flow and flow patterns in relation to functional recovery measured by NIHSS and modified Rankin Scale (mRS) scores.

DETAILED DESCRIPTION:
TRADE-AIS (Transcranial Doppler Evaluation - Acute Ischemic Stroke) is a prospective, single-center, observational cohort study designed to evaluate the prognostic value of transcranial Doppler ultrasound (TCD) in patients with acute ischemic stroke (AIS). The study will be conducted at Clínica México, a secondary-level hospital located in Piedras Negras, Coahuila, Mexico.

Upon presentation to the emergency department or inpatient stroke unit, patients diagnosed with AIS will undergo a baseline neurological examination, including NIH Stroke Scale (NIHSS) scoring. A transcranial Doppler ultrasound will then be performed within 24 hours of symptom onset. The TCD protocol will include insonation of the middle cerebral arteries (MCAs), anterior and posterior communicating arteries, and basilar artery, using a 2-MHz probe via the temporal window.

Parameters to be recorded include:

Mean flow velocity (Vm) in the MCA

Pulsatility index (PI)

Presence and pattern of collateral flow (e.g., via anterior communicating artery)

Abnormal waveforms such as reverberant, absent, or blunted flow

Patients will be clinically monitored throughout their hospital stay. Follow-up NIHSS scoring will be conducted at 72 hours. Functional status at discharge will be assessed using the modified Rankin Scale (mRS). The primary aim is to correlate early hemodynamic findings with short-term neurological evolution. Secondary aims include assessing the association of collateral circulation with clinical improvement and determining whether TCD-derived indices can serve as non-invasive prognostic markers.

All diagnostic and therapeutic decisions (e.g., reperfusion therapy, ICU admission) will be made by the attending medical team independently of study procedures. No experimental interventions are included.

The study intends to demonstrate that early bedside neurosonology can provide clinically relevant prognostic information, particularly useful in settings with limited access to advanced imaging modalities like CT perfusion or MRI.

Data will be collected and managed using encrypted case report forms. Statistical analysis will include correlation tests and multivariate regression models to adjust for clinical covariates.

The primary outcome is the correlation between baseline MCA flow velocity and the change in NIHSS score at 72 hours. Secondary outcomes include:

The association between collateral circulation and clinical improvement,

Functional status at hospital discharge, assessed using the modified Rankin Scale (mRS).

The study will take place over 12 months at Clínica México, a secondary-level hospital located in Piedras Negras, Coahuila, Mexico. The study is non-interventional: all treatment decisions, including eligibility for thrombolysis or endovascular therapy, are made by the attending clinical team and are not influenced by study participation.

This investigation is designed to assess the prognostic value of TCD as a non-invasive, bedside tool for early risk stratification in AIS, particularly in settings with limited access to advanced neuroimaging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical diagnosis of acute ischemic stroke
* Onset of symptoms ≤ 24 hours before admission
* Underwent or will undergo transcranial Doppler ultrasound within 24 hours of symptom onset
* Able to provide informed consent or consent obtained from a legal representative

Exclusion Criteria:

* Evidence of intracerebral hemorrhage on imaging
* Inadequate temporal acoustic window for transcranial Doppler
* Intubated or hemodynamically unstable prior to Doppler evaluation
* Known diagnosis of neurodegenerative disease significantly affecting baseline neurological function (e.g., advanced dementia, Parkinson's disease)
* Refusal to participate or withdrawal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in NIHSS score from baseline to 72 hours | 72 hours
  Neurological status will be assessed using the National Institutes of Health Stroke Scale (NIHSS) at baseline (upon admission) and again at 72 hours. The primary objective is to evaluate the correlation between initial transcranial Doppler (TCD) measurements-specifically, mean flow velocity and pulsatility index in the middle cerebral artery-and the degree of clinical improvement or deterioration, as reflected by changes in NIHSS score. A greater reduction in NIHSS score indicates better neurological recovery.
  The NIH Stroke Scale (NIHSS) is a standardized, 15-item clinical assessment tool used to evaluate the severity of neurologic deficits in patients with acute stroke. The total NIHSS score ranges from 0 to 42, where:
  0 = no stroke symptoms
  Higher scores indicate greater stroke severity and worse neurological outcomes
  The scale includes assessments of level of consciousness, gaze, visual fields, motor strength, limb ataxia, sensory function, language, and neglect.

SECONDARY OUTCOMES:
Presence of collateral circulation associated with ≥ 4-point NIHSS improvement | 7 days
  Collateral circulation will be assessed using transcranial Doppler ultrasound within 24 hours of symptom onset. Collaterals will be defined as the presence of cross-flow or increased velocity in the anterior or posterior communicating arteries. Clinical improvement is defined as a reduction of ≥4 points on the NIHSS score from baseline to day 7. The association between collateral flow and neurological improvement will be analyzed.
  The NIH Stroke Scale (NIHSS) is a standardized, 15-item clinical assessment tool used to evaluate the severity of neurologic deficits in patients with acute stroke. The total NIHSS score ranges from 0 to 42, where:
  0 = no stroke symptoms
  Higher scores indicate greater stroke severity and worse neurological outcomes
  The scale includes assessments of level of consciousness, gaze, visual fields, motor strength, limb ataxia, sensory function, language, and neglect.
Functional status at discharge (modified Rankin Scale) | At hospital discharge (within 14 days of admission)
  The patient's functional outcome will be assessed at discharge using the modified Rankin Scale (mRS), which ranges from 0 (no symptoms) to 6 (death). The distribution of mRS scores will be analyzed in relation to transcranial Doppler findings, including mean flow velocity, pulsatility index, and flow pattern, to determine their prognostic significance.

IPD SHARING:
Plan to Share IPD: Undecided
Not decided.

REFERENCES:
- [Background] Alexandrov AV, Sloan MA, Wong LK, Douville C, Razumovsky AY, Koroshetz WJ, Kaps M, Tegeler CH; American Society of Neuroimaging Practice Guidelines Committee. Practice standards for transcranial Doppler ultrasound: part I--test performance. J Neuroimaging. 2007 Jan;17(1):11-8. doi: 10.1111/j.1552-6569.2006.00088.x. PMID 17238867